CLINICAL TRIAL: NCT00642603
Title: A Randomized, Open Label Study of the Effect of First Line Treatment With Xeloda in Combination With Avastin and Either Short Course Irinotecan or Short Course Oxaliplatin on Progression-free Survival in Patients With Metastatic Colorectal Cancer
Brief Title: A Study of Xeloda (Capecitabine) in Combination With Avastin + Short Course Chemotherapy in Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21567
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Bevacizumab; Oxaliplatin; Irinotecan

ARMS (2):
- XELOX + bevacizumab (Q2W) (Experimental)
  Interventions: Drug: capecitabine [Xeloda]; Drug: bevacizumab [Avastin]; Drug: oxaliplatin
- XELIRI + bevacizumab (Q2W) (Experimental)
  Interventions: Drug: capecitabine [Xeloda]; Drug: bevacizumab [Avastin]; Drug: irinotecan

INTERVENTIONS:
Drug: capecitabine [Xeloda] — 1000 mg/m2 twice-daily, taken orally on Days 1-7 of each 2 week cycle
  Arms: XELOX + bevacizumab (Q2W)
Drug: capecitabine [Xeloda] — 1000 mg/m2 twice-daily, taken orally on Days 1-7 of each 2 week cycle
  Arms: XELIRI + bevacizumab (Q2W)
Drug: bevacizumab [Avastin] — 5 mg/kg taken intravenously on Day 1 of each 2 week cycle
Drug: oxaliplatin — 85 mg/m2 taken intravenously on Day 1 of each 2 week cycle, for first 9 cycles
  Arms: XELOX + bevacizumab (Q2W)
Drug: irinotecan — 135 mg/m2 taken intravenously on Day 1 of each 2 week cycle, for first 9 cycles
  Arms: XELIRI + bevacizumab (Q2W)

SUMMARY:
This 2-arm study was designed to evaluate the efficacy and safety of 2 treatment regimens of Xeloda and Avastin, with either irinotecan or oxaliplatin administered for the first 12 cycles, as first line treatment in patients with metastatic colorectal cancer. Patients were randomized to receive 2-weekly cycles of treatment with either: 1) Xeloda, Avastin and oxaliplatin; or 2) Xeloda, Avastin and irinotecan. After 9 cycles, patients continued to receive maintenance treatment with Xeloda + Avastin. The anticipated time on study treatment was until disease progression, and the target sample size was 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years of age
* Histologically confirmed adenocarcinoma of colon or rectum, with unresectable metastatic or locally advanced disease
* ≥1 measurable target lesion
* Ambulatory, with an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1

Exclusion Criteria:

* Prior systemic therapy for advanced or metastatic disease
* History of another malignancy within last 5 years, except cured basal cell cancer of skin or cured cancer in situ of the cervix
* Clinically significant cardiovascular disease
* Current or recent use of full dose oral warfarin or full dose parenteral anticoagulants or thrombolytic agents
* Chronic daily treatment with >325 mg/day aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (71):
- United States (71):
  - PARK Springs, Arizona
  - Sedona, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Colton, California
  - Greenbrae, California
  - Loma Linda, California
  - Modesto, California
  - Montebello, California
  - Pomona, California
  - Sacramento, California
  - Norwich, Connecticut
  - Waterbury, Connecticut
  - Lake Worth, Florida
  - Miami Shores, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Ocoee, Florida
  - Marietta, Georgia
  - Niles, Illinois
  - Paducah, Kentucky
  - Alexandria, Louisiana
  - Baltimore, Maryland
  - Westminster, Maryland
  - Pittsfield, Massachusetts
  - Worcester, Massachusetts
  - Kalamazoo, Michigan
  - Duluth, Minnesota
  - Jefferson City, Missouri
  - Great Falls, Montana
  - Las Vegas, Nevada
  - Neptune City, New Jersey
  - Albuquerque, New Mexico
  - Santa Fe, New Mexico
  - Brooklyn, New York
  - Huntington Station, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Canton, Ohio
  - Eugene, Oregon
  - Ephrata, Pennsylvania
  - Langhorne, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scranton, Pennsylvania
  - Charleston, South Carolina
  - Florence, South Carolina
  - Sumter, South Carolina
  - Chattanooga, Tennessee
  - Cookeville, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Arlington, Texas
  - Beaumont, Texas
  - Bedford, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Garland, Texas
  - Lewisville, Texas
  - Mesquite, Texas
  - Paris, Texas
  - Round Rock, Texas
  - San Antonio, Texas
  - Southlake, Texas
  - Sugar Land, Texas
  - Waco, Texas
  - Webster, Texas
  - Salt Lake City, Utah
  - Christiansburg, Virginia
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- XELOX + Bevacizumab (Q2W): Capecitabine orally at a dose of 1000 mg/m2 twice daily, bevacizumab intravenously at a dose of 5 mg/kg on Day 1 of each cylce, and oxaliplatin intravenously at a dose of 85 mg/m2 on Day 1 following bevacizumab for the first 12 cycles only. Each cycle is 14 days consisting of 7 days of treatment followed by 7 days without treatment.
- XELIRI + Bevacizumab (Q2W): Capecitabine orally at a dose of 1000 mg/m2 twice daily, bevacizumab intravenously at a dose of 5 mg/kg on Day 1 of each cycle, and irinotecan intravenously at a dose of 135 mg/m2 on Day 1 following bevacizumab for the first 12 cycles only. Each cycle is 14 days consisting of 7 days of treatment followed by 7 days without treatment.
Period: Overall Study
Arm/Group | XELOX + Bevacizumab (Q2W) | XELIRI + Bevacizumab (Q2W)
Started | 21 | 20
Safety Population | 19 | 20
Completed | 0 | 2
Not Completed | 21 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XELOX + Bevacizumab (Q2W) | XELIRI + Bevacizumab (Q2W) | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (12.06) | 60.6 (9.89) | 62.3 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) in U.S. Patients Only
Description: PFS was defined as the time from the date of randomization to the first documented occurrence of disease progression or death due to any cause.
Time Frame: From first patient enrolled up to approximately 48 months
Population: This study was terminated early because interim data from a predecessor study invalidated the scientific rationale that provided justification for the conduct of this study. Efficacy analyses were not performed.
Arm/Group | XELOX + Bevacizumab (Q2W) | XELIRI + Bevacizumab (Q2W)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Safety analysis population = received at least one dose of study medication. Note: The incidence of each AE/SAE is reported as the number of participants experiencing the event, not the number of occurrences for each AE/SAE.
Arm/Group | XELOX + Bevacizumab (Q2W) | XELIRI + Bevacizumab (Q2W)
Serious Adverse Events (participants affected / at risk) | 4/19 | 7/20
Other Adverse Events (participants affected / at risk) | 17/19 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XELOX + Bevacizumab (Q2W) (N=19) | XELIRI + Bevacizumab (Q2W) (N=20)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Hypertrophic Cardiomyopathy (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lacunar Infarction (Nervous system disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XELOX + Bevacizumab (Q2W) (N=19) | XELIRI + Bevacizumab (Q2W) (N=20)
Diarrhoea (Gastrointestinal disorders) | 9 | 11
Nausea (Gastrointestinal disorders) | 6 | 11
Vomiting (Gastrointestinal disorders) | 4 | 5
Abdominal Pain (Gastrointestinal disorders) | 1 | 6
Constipation (Gastrointestinal disorders) | 3 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 2
Oral Pain (Gastrointestinal disorders) | 0 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Anal Pruritus (Gastrointestinal disorders) | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 7 | 7
Pyrexia (General disorders) | 1 | 3
Asthenia (General disorders) | 0 | 3
Malaise (General disorders) | 1 | 2
Catheter Related Complication (General disorders) | 0 | 1
Catheter Thrombosis (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Gait Disturbance (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0
Infusion Related Reaction (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Temperature Intolerance (General disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 9 | 0
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1
Burning Sensation (Nervous system disorders) | 0 | 1
Disturbance In Attention (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Livedo Reticularis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Anorexia (Metabolism and nutrition disorders) | 5 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2
Food Intolerance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysaesthesia Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 0 | 2
Abscess Intestinal (Infections and infestations) | 1 | 0
Clostridial Infection (Infections and infestations) | 0 | 1
Clostridium Bacteraemia (Infections and infestations) | 1 | 0
Escherichia Bacteraemia (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Weight Decreased (Investigations) | 1 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Sputum Abnormal (Investigations) | 1 | 0
X-ray Abnormal (Investigations) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Flushing (Vascular disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0
Tooth Extraction (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early because interim data from a predecessor study invalidated the scientific rationale that provided justification for the conduct of this study. Efficacy analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.